CLINICAL TRIAL: NCT01184508
Title: A Randomized, Double-Blind, Placebo Controlled Proof of Concept Study of LY2300559 in Patients With Migraine
Brief Title: A Study in Migraine Prevention
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Elevation of ALT and AST in some patients.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13313; I1N-MC-CDBE (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Migraine Headache
Keywords: classic with aura; common without aura; migraine; headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — LY2300559

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2300559 (Experimental)
  Interventions: Drug: LY2300559
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Administered orally, once daily, for 12 weeks
  Arms: Placebo
Drug: LY2300559 — 300 milligrams (mg) administered orally, once daily, for 12 weeks
  Arms: LY2300559

SUMMARY:
The primary objective of this study is to measure the change in frequency of migraine attacks per 28 days in migraine patients being treated orally with LY2300559 for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Are migraine patients with migraine onset before 50 years of age
* Present with diagnosis of at least 1 year with migraine attack defined by International Headache Society (IHS) guidelines
* Have a frequency of 4 to 14 migraine attacks, with or without aura, per month (with no more than 14 headache days per month, migraine or non-migraine) for at least the last 6 months
* Female patients of childbearing potential must test negative for pregnancy at the time of enrollment and agree to use a reliable method of birth control during the study

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the previous 6 months from a migraine clinical trial involving an investigational drug or device or off-label use of a drug or device
* Are currently enrolled in, or discontinued within the previous 30 days from screening from a non-migraine clinical trial involving an investigational drug or device or off-label use of a drug or device, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have previously completed or withdrawn from this study or any other study investigating LY2300559
* Have known allergies to LY2300559 or related compounds (such as montelukast)
* Are under treatment with medication or procedures for prevention of migraine, or are taking any other medications that are excluded by the protocol
* Have a history of alcohol or drug abuse/dependence within the past 3 months of screening or are currently using alcohol, drugs of abuse (including opioids, barbiturates, and marijuana), or any prescribed or over-the-counter medication in a manner that the investigator considers indicative of abuse/dependence
* Screen positive for drugs of abuse
* Patients with medication overuse headache as per IHS definition
* Have a body mass index (BMI) of less than 18.5 or greater than or equal to 35.0
* Have history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, constituting a risk when taking the study medication or interfering with the interpretation of the data
* Show evidence of serious active neuropsychiatric disease including, but not limited to, bipolar disorder, schizophrenia, psychosis, cluster B personality disorders [for example (eg), borderline personality disorder or narcissistic personality disorder], obsessive-compulsive disorder, or other serious mood, anxiety, depression, or substance/alcohol use disorders
* Have ever in his/her lifetime attempted suicide, have any recent suicidal ideation within the last 3 months, or are at significant risk to commit suicide, as judged by the investigator
* Show evidence or have history of neurological disease such as cerebral vascular accident, pseudotumor cerebri, multiple sclerosis, transient ischemic attack, syncopal episodes, encephalitis, or meningitis
* Have a history or seizures other than febrile
* Female patients who are pregnant or breast-feeding
* Females of childbearing potential who are not using a clinically acceptable method of birth control (eg, oral contraceptives or abstinence)
* Are unwilling or unable to comply with the use of a data collection device to directly record patient data
* Are otherwise unable to comply with the requirements of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- United States (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Long Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fairfield, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to randomization, participants completed screening and washout followed by a 28-day baseline period to determine the number of migraine attacks participants experienced without the use of preventative medications. Participant Flow and results based on participants, post-randomization (12-week treatment and 4-week follow-up periods combined).
Groups:
- Placebo: Capsules administered orally, once daily, for 12 weeks.
- LY2300559: 300 milligrams (mg) administered orally as two 150-mg capsules, once daily, for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | LY2300559
Started | 45 | 42
Received at Least 1 Dose of Study Drug | 45 | 41
Completed | 29 | 27
Not Completed | 16 | 15
Not completed — Adverse Event | 4 | 6
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Protocol Violation | 3 | 1
Not completed — Sponsor Decision | 5 | 2
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Randomized, Not Treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat 1 (mITT1) population: participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | LY2300559 | Total
Number analyzed (Participants) | 45 | 41 | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (10.09) | 41.4 (12.17) | 42.4 (11.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 33 | 71
  Male | 7 | 8 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 3 | 3
  Black or African American | 2 | 5 | 7
  Multiple | 1 | 1 | 2
  White | 42 | 32 | 74
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 41 | 86
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] — BMI is an estimate of body fat based on body weight divided by height squared.
  kilograms per square meter (kg/m^2) | 26.5 (3.65) | 26.3 (5.13) | 26.4 (4.39)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12 Week Endpoint in the Number of Migraine Attacks
Description: The definition of a migraine (a headache lasting 4 to 72 hours) was based on the International Headache Society (IHS) diagnostic criteria. The number of migraine attacks per month was normalized to a 28-day month and calculated as the (number of migraine attacks*28 days)/number of days in the specified month.
Time Frame: Baseline and Month 3
Population: Randomized participants (pts) who had at least 4 migraines and/or probable migraine headaches during the baseline period, who received at least 1 dose of study drug, and for whom had at least 1 post-randomization efficacy data for the specified endpoint was available.
Measure: Mean (Standard Deviation); unit: migraine attacks
Arm/Group | Placebo | LY2300559
Number analyzed (Participants) | 31 | 33
migraine attacks
  Baseline | 5.2 (1.03) | 5.5 (1.50)
  Month 3: number analyzed (Participants) | 21 | 22
  Month 3 | 3.4 (1.88) | 2.8 (2.08)
Statistical Analysis 1: Comparison: Placebo vs LY2300559; Test type: Superiority or Other; p = 0.085, Mixed-effects model repeated-measures — The comparison between LY2300559 and placebo for the LS mean change from baseline to Month 3 in the number of migraine attacks was conducted at a 2-sided alpha level of 0.10 without adjustment for multiplicity; Fixed effects: pooled investigator, treatment (tx) group, month, tx group*month, baseline, baseline*month; Random effect: pts; Repeated effect: month; Least squares (LS) mean difference (Net) = -1.03, 90% CI 2-sided [-2.02 to -0.05]

2. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Severity of Migraine Intensity (Mild, Moderate, Severe)
Description: The participant-reported severity of migraines was rated on a 3-point categorical scale (Mild, Moderate, or Severe). Participants could report a severity of none (score = 0), mild (1), moderate (2), or severe (3). In general, if a headache was mild, daily activities could be resumed and little to no medication was taken. Moderate headaches required medication and effected daily activities. Severe headaches were debilitating and required medication. If a participant had multiple migraines during Month 3 (normalized to 28 days), the most severe migraine was analyzed.
Time Frame: Baseline and Month 3
Population: Randomized participants who had at least 4 migraines and/or probable migraine headaches during the baseline period, who received at least 1 dose of study drug, and for whom at least 1 post-randomization efficacy data for the specified endpoint was available.
Measure: Number; unit: participants
Arm/Group | Placebo | LY2300559
Number analyzed (Participants) | 31 | 33
participants
  Mild, Baseline | 0 | 0
  Mild, Month 3 | 3 | 0
  Moderate, Baseline | 8 | 12
  Moderate, Month 3 | 7 | 14
  Severe, Baseline | 23 | 21
  Severe, Month 3 | 10 | 4

3. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Average Duration of Migraine Symptoms
Description: The duration of migraine symptoms was the amount of time from the beginning of each individual migraine attack to the end of each migraine attack. Two attacks separated by <24 hours were considered part of the same migraine and duration was calculated as such. Migraine symptoms included photophobia, phonophobia, nausea, and vomiting. No data collected for aura and vomiting's migraine symptoms.
Time Frame: Baseline and Month 3
Population: Randomized participants (pts) who had at least 4 migraines/probable migraines during the baseline period, who received at least 1 dose of study drug, and had at least 1 post-randomization efficacy data for the specified endpoint.No data collected for aura and vomiting's migraine symptoms.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Placebo | LY2300559
Number analyzed (Participants) | 31 | 31
hours
  Duration of Photophobia, Baseline | 15.3 (12.75) | 18.3 (12.70)
  Duration of Photophobia, Month 3: number analyzed (Participants) | 16 | 15
  Duration of Photophobia, Month 3 | 16.3 (19.80) | 18.7 (13.87)
  Duration of Phonophobia, Baseline | 15.7 (10.59) | 16.4 (12.54)
  Duration of Phonophobia, Month 3: number analyzed (Participants) | 15 | 14
  Duration of Phonophobia, Month 3 | 17.1 (19.98) | 17.4 (11.19)
  Duration of Nausea, Baseline: number analyzed (Participants) | 27 | 25
  Duration of Nausea, Baseline | 12.8 (12.15) | 13.9 (17.61)
  Duration of Nausea, Month 3: number analyzed (Participants) | 15 | 10
  Duration of Nausea, Month 3 | 17.5 (16.26) | 14.1 (10.42)
Statistical Analysis 1: Comparison: Placebo vs LY2300559; Test type: Superiority or Other; p = 0.770, Mixed-effects model repeated-measures — The p-value is for the change from baseline to Month 3 in average duration of photophobia; [statistical method as in outcome 1, analysis 1]; Least squares (LS) mean difference = 1.75, 90% CI 2-sided [-8.27 to 11.76]
Statistical Analysis 2: Comparison: Placebo vs LY2300559; Test type: Superiority or Other; p = 0.276, Mixed-effects model repeated-measures — The p-value is for the change from baseline to Month 3 in average duration of phonophobia; Fixed effects: pooled investigator, tx group, month, tx group*month, baseline, baseline*month; Random effect: pts; Repeated effect: month; LS mean difference = 7.30, 90% CI 2-sided [-3.91 to 18.52]
Statistical Analysis 3: Comparison: Placebo vs LY2300559; Test type: Superiority or Other; p = 0.606, Mixed-effects model repeated-measures — The p-value is for the change from baseline to Month 3 in average duration of nausea; [statistical method as in outcome 3, analysis 2]; LS mean difference = -2.70, 90% CI 2-sided [-11.51 to 6.10]

4. Secondary Outcome: Mean Change From Baseline to 12 Week Endpoint in the Number of Migraine Days
Description: A migraine day was any day with a migraine attack (a headache lasting 4 to 72 hours). The number of migraine days per month was normalized to a 28-day month and calculated as the (number of migraine days*28)/number of days in the specified month.
Time Frame: Baseline and Month 3
Population: Randomized participants (pts) who had at least 4 migraines and/or probable migraine headaches during the baseline period, who received at least 1 dose of study drug, and for whom at least 1 post-randomization efficacy data for the specified endpoint was available.
Measure: Mean (Standard Deviation); unit: migraine days
Arm/Group | Placebo | LY2300559
Number analyzed (Participants) | 31 | 33
migraine days
  Baseline | 8.8 (2.56) | 10.5 (4.47)
  Month 3: number analyzed (Participants) | 21 | 22
  Month 3 | 6.3 (3.77) | 4.9 (3.80)
Statistical Analysis 1: Comparison: Placebo vs LY2300559; Test type: Superiority or Other; p = 0.174, Mixed-effects model repeated-measures — The p-value is for the mean change from baseline to Month 3 in the number of migraine days; [statistical method as in outcome 1, analysis 1]; Least squares (LS) mean difference = -1.57, 90% CI 2-sided [-3.48 to 0.34]

5. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Clinical Global Impression of Improvement (CGI-I)
Description: The CGI-I was a 1-item scale that measured the clinician's perception of the improvement in migraine symptoms compared with the start of treatment. Scores ranged from 1 (very much improved) to 7 (very much worse). A score of 4 indicated no change.
Time Frame: Baseline(Day 28) and Week 12 (Day 84)
Population: Randomized participants who had at least 4 migraines and/or probable migraine headaches during the baseline period, who received at least 1 dose of study drug and, for whom at least 1 post-randomization efficacy data for the specified endpoint was available.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo | LY2300559
Number analyzed (Participants) | 31 | 33
units on a scale
  Baseline | 4.0 [4.0 to 4.0] | 4.0 [3.0 to 5.0]
  Week 12: number analyzed (Participants) | 20 | 25
  Week 12 | 3.0 [1.0 to 5.0] | 2.0 [1.0 to 5.0]

6. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Patient's Global Impression of Improvement (PGI-I)
Description: The PGI-I was a 1-item scale that measured the participant's perception of improvement in migraine symptoms compared with the start of treatment. Scores ranged from 1 (very much improved) to 7 (very much worse). A score of 4 indicated no change.
Time Frame: Baseline (Day 28) and Week 12 (Day 84)
Population: as for outcome 2
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo | LY2300559
Number analyzed (Participants) | 31 | 33
units on a scale
  Baseline | 4.0 [4.0 to 5.0] | 4.0 [3.0 to 5.0]
  Week 12: number analyzed (Participants) | 20 | 25
  Week 12 | 2.5 [1.0 to 5.0] | 2.0 [1.0 to 5.0]

7. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Migraine-Specific Quality of Life Questionnaire (MSQ) Score
Description: The MSQ was a 14-item self-administered scale that assessed the participant's perception of quality of life for 3 dimensions [role restriction or restrictive function (Items 1-7), role prevention or preventive function (Items 8-11), and emotional function (Items 12-14)]. Participants rated each item from 1 (none of the time) to 6 (all of the time). Since each item was presented as a negative statement, participant responses were recoded before item scores were calculated. Then, dimension scores were calculated as the sum of the recoded items for that specific dimension. Each dimension score was transformed into a score that ranged from 0 to 100. The transformation formula for the restrictive function = [(dimension score-7)*100]/35, for the preventive function = [(dimension score-4)*100]/20, and for the emotional function = [(dimension score-3)*100]/15. A lower score indicated a poorer quality of life associated with that domain.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | LY2300559
Number analyzed (Participants) | 31 | 33
units on a scale
  Restrictive Function Score, Baseline | 62.8 (15.20) | 59.0 (17.71)
  Restrictive Function Score, Week 12: number analyzed (Participants) | 20 | 25
  Restrictive Function Score, Week 12 | 74.6 (18.44) | 80.1 (15.62)
  Preventive Function Score, Baseline | 79.0 (16.09) | 76.4 (20.24)
  Preventive Function Score, Week 12: number analyzed (Participants) | 20 | 25
  Preventive Function Score, Week 12 | 85.5 (17.08) | 89.4 (11.49)
  Emotional Function Score, Baseline | 70.8 (20.20) | 70.3 (26.83)
  Emotional Function Score, Week 12: number analyzed (Participants) | 20 | 25
  Emotional Function Score, Week 12 | 84.7 (19.24) | 88.0 (14.40)
Statistical Analysis 1: Comparison: Placebo vs LY2300559; Test type: Superiority or Other; p = 0.963, ANCOVA — The p-value is for the change from baseline to Week 12 in MSQ restrictive function score; Fixed effects: investigator (pooled site), treatment group, visit, treatment group*visit, baseline and baseline*visit; Least squares (LS) mean difference = -0.27, 90% CI 2-sided [-9.76 to 9.23]
Statistical Analysis 2: Comparison: Placebo vs LY2300559; Test type: Superiority or Other; p = 0.591, ANCOVA — The p-value is for the change from baseline to Week 12 in MSQ preventive function score; Fixed effects: investigator (pooled site), treatment group, visit, treatment group*visit, baseline and baseline*visit; LS mean difference = -2.17, 90% CI 2-sided [-8.85 to 4.50]
Statistical Analysis 3: Comparison: Placebo vs LY2300559; Test type: Superiority or Other; p = 0.720, ANCOVA — The p-value is for the change from baseline to Week 12 in MSQ emotional function score; Fixed effects: investigator (pooled site), treatment group, visit, treatment group*visit, baseline and baseline*visit; LS mean difference = 1.89, 90% CI 2-sided [-6.81 to 10.58]

8. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Migraine Interictal Burden Scale (MIBS-4) Overall Weighted Score
Description: MIBS-4 was a 4-item self-administered scale that assessed the impact of headaches on the participant's life between headache attacks. Each item measured a specific domain (impairment in work or school, impairment in family and social life, difficulty making plans or commitments, or emotional/affective and cognitive distress). For each item and domain, scores were weighted as follows: Don't know (0), Never (0), Rarely (1), Some of the time (2), Much of the time (3), and All of the time (4). The overall weighted score was the sum of the domain scores and ranged from 0 to 16. Higher scores indicated a greater impact of headaches on the participant's life between headache attacks.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | LY2300559
Number analyzed (Participants) | 31 | 33
units on a scale
  Baseline | 4.0 (3.72) | 3.0 (3.21)
  Week 12: number analyzed (Participants) | 20 | 25
  Week 12 | 2.3 (3.15) | 2.1 (2.34)
Statistical Analysis 1: Comparison: Placebo vs LY2300559; Test type: Superiority or Other; p = 0.688, ANCOVA — The p-value is for the change from baseline to Week 12 in MIBS-4 overall weighted score; Fixed effects: pooled investigator, treatment group, and baseline; Least squares (LS) mean difference = -0.25, 90% CI 2-sided [-1.30 to 0.80]

9. Secondary Outcome: Pharmacokinetics: Area Under the Plasma Concentration-Time Curve at the Steady State (AUCtau,ss) of LY2300559
Time Frame: Baseline and Week 8 (1 to 3 hours postdose), Weeks 2 and 4 (predose and 1 to 3 hours postdose), Week 12 (predose, 1 to 3 hours postdose, and 5 hours postdose)
Population: Participants who received at least 1 dose of study drug and had at least 1 evaluable pharmacokinetic sample.
Measure: Median (95% Confidence Interval); unit: nanogram*hours per milliliter (ng*h/mL)
Arm/Group | LY2300559
Number analyzed (Participants) | 41
nanogram*hours per milliliter (ng*h/mL) | 479000 [131000 to 1156000]

10. Secondary Outcome: Percentage of Participants Using Breakthrough Medications
Description: Participants were allowed to use a pre-approved list of medications for the treatment of breakthrough migraines during the study, as long as the treatments were the same as those used and reported during the baseline period. Any medications or procedures to prevent migraines were not allowed. Percentage of participants = (number of participants using breakthrough medication/total number of participants)*100. Each month was normalized to a 28-day month.
Time Frame: Month 3
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | LY2300559
Number analyzed (Participants) | 21 | 22
percentage of participants | 95.2 | 86.4
Statistical Analysis 1: Comparison: Placebo vs LY2300559; Test type: Superiority or Other; p = 0.607, Fisher Exact — The p-value is for the percentage of participants using breakthrough medication at Month 3

11. Other Pre Specified Outcome: Change From Baseline to 12 Week Endpoint in Breakthrough Treatment Therapy for Acute Migraine Attacks
Description: Participants were allowed to use a pre-approved list of medications for the treatment of breakthrough migraines during the study, as long as the treatments were the same as those used and reported during the baseline period. Any medications or procedures to prevent migraines were not allowed. The mean number was calculated by the breakthrough (BH) medications (meds) per migraine used by each participant per month. Each month was normalized to a 28-day month.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: BH meds/migraine by participants/month
Arm/Group | Placebo | LY2300559
Number analyzed (Participants) | 19 | 17
BH meds/migraine by participants/month | 0.34 (0.6) | -0.03 (0.6)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 16
Arm/Group | Placebo | LY2300559
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/41
Other Adverse Events (participants affected / at risk) | 32/45 | 30/41
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=45) | LY2300559 (N=41)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (5) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 5 (5) | 7 (7)
Feeling abnormal (General disorders) | 2 (2) | 0 (0)
Therapeutic response unexpected (General disorders) | 2 (2) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 8 (8)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 8 (8)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 2 (2)
Weight increased (Investigations) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 5 (6) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was stopped due to clinically significant elevations of alanine aminotransferase (ALT) and aspartate aminotransferase (AST) in some participants. Due to early study termination, the planned sample size was not met.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days